CLINICAL TRIAL: NCT01293552
Title: Clinical Trial To Evaluate Botulinum Neurotoxin Type A (ANT-1207) In Subjects With Acne
Brief Title: Clinical Trial To Evaluate ANT-1207 In Subjects With Acne
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Anterios Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ANT-1207-101-ACNE
Record Dates: First submitted 2011-02-09; First posted 2011-02-10 (Estimated); Last update posted 2013-07-04 (Estimated); Status verified 2013-06

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Control (Placebo Comparator): blank vehicle formulation
  Interventions: Biological: Vehicle
- Dose 1 (Experimental): Dose 1
  Interventions: Biological: ANT-1207
- Dose 2 (Experimental): Dose 2
  Interventions: Biological: ANT-1207
- Dose 3 (Experimental): Dose 3
  Interventions: Biological: ANT-1207
- Dose 4 (Experimental): Dose 4
  Interventions: Biological: ANT-1207

INTERVENTIONS:
Biological: ANT-1207 — single dose application
  Arms: Dose 1; Dose 2; Dose 3; Dose 4
Biological: Vehicle
  Other Names: Placebo
  Arms: Control

SUMMARY:
The purpose of this study is to provide evidence of the safety, tolerance, and efficacy of ANT-1207 in the treatment of acne.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of moderate to severe facial acne
* 15 to 40 papules and pustules, and 5 to 50 open and/or closed comedones
* no presence of nodules
* female subjects must be not pregnant and non-lactating

Exclusion Criteria:

* presence of 1 or more nodules
* use of topical steroids on the face 4 weeks prior and during the study
* use of systemic corticosteroids 6 weeks prior and during the study
* topical or systemic acne treatment in the 4 weeks prior to Baseline

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2011-01; Primary Completion 2012-04 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Efficacy will be assessed by lesion count. | Week 4
  inflammatory lesion count (papules, pustules, and nodules) and non-inflammatory lesion count (open and closed comedones)

SECONDARY OUTCOMES:
Change from Baseline in Investigator Global Assessment Score | Week 1, 2, 4, 8, and 12
Change from Baseline in Lesion Count | Week 1, 2, 4, 8, 12

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Total Skin & Beauty Dermatology Center, Birmingham, Alabama
  - International Dermatology Research, Miami, Florida
  - Palm Beach Esthetic Dermatology and Laser Center, West Palm Beach, Florida
  - Gwinnett Clinical Research Center Inc., Snellville, Georgia
  - Dermatology Specialists Research, LLC, Louisville, Kentucky
  - William Coleman III, MD, APMC, Metairie, Louisiana
  - Grekin Skin Institute, Warren, Michigan
  - The Dermatology Group, P.C., Verona, New Jersey
  - Gramercy Park Dermatology, New York, New York
  - Skin Search of Rochester, Inc, Rochester, New York
  - Dermatology Consulting Services, High Point, North Carolina
  - Penn State Hershey Medical Center Department of Dermatology, Hershey, Pennsylvania
  - Yardley Dermatology Associates, Yardley, Pennsylvania
  - The Skin Wellness Center, Knoxville, Tennessee
  - DermResearch, Inc., Austin, Texas